CLINICAL TRIAL: NCT07214558
Title: he Effect of Spinal and General Anesthesia on Inflammatory Response Measured by Delta Neutrophil Index in Patients Undergoing Total Knee Arthroplasty: A Prospective Observational Study
Brief Title: Spinal Versus General Anesthesia and Inflammatory Response Measured by Delta Neutrophil Index in Total Knee Arthroplasty: An Observational Study
Acronym: DNA-TKA
Status: Completed | Type: Observational
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Principal Investigator, Sevim Şenol Karataş, Principal Investigator, Elazıg Fethi Sekin Sehir Hastanesi
Other Study IDs: EFSH-ANES-2025-09-DELTANEUTROP
Record Dates: First submitted 2025-09-22; First posted 2025-10-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Response in Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Spinal Anesthesia; General Anesthesia; Delta Neutrophil Index; Inflammatory Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal Anesthesia Group: Patients undergoing total knee arthroplasty under spinal anesthesia. The choice of anesthesia is based on clinical decision-making in routine practice.
  Interventions: Other: Routine Clinical Anesthesia Practice
- General Anesthesia Group: Patients undergoing total knee arthroplasty under general anesthesia. The choice of anesthesia is based on clinical decision-making in routine practice.
  Interventions: Other: Routine Clinical Anesthesia Practice

INTERVENTIONS:
Other: Routine Clinical Anesthesia Practice — Patients undergoing total knee arthroplasty will receive either spinal or general anesthesia as determined by routine clinical practice and the attending anesthesiologist's decision. Investigators will not influence the choice of anesthesia method.

SUMMARY:
This study aims to compare the effects of spinal versus general anesthesia on the inflammatory response measured by Delta Neutrophil Index (DNI) in patients undergoing total knee arthroplasty. The study is prospective and observational. A total of at least 84 patients will be included, with anesthesia type determined according to routine clinical practice. Preoperative and postoperative blood tests will be analyzed, and no additional blood samples will be required.

DETAILED DESCRIPTION:
This prospective observational study will be conducted at Elazig Fethi Sekin City Hospital, Department of Anesthesiology and Reanimation. Patients undergoing total knee arthroplasty will be assigned to two groups based on the anesthesia method used in routine practice: spinal anesthesia or general anesthesia. The primary outcome measure is the Delta Neutrophil Index (DNI), an inflammation marker automatically calculated by hematology analyzers using complete blood count parameters. DNI values will be compared preoperatively and postoperatively between groups. Additional data including age, sex, ASA classification, duration of surgery, hemogram parameters, and perioperative complications will be collected. The sample size calculation indicated that a minimum of 42 patients per group (total 84) are required to detect significant differences in DNI levels with 80% power at a 5% significance level. Statistical analyses will include Kolmogorov-Smirnov test for normality, independent t test or Mann-Whitney U test for between-group comparisons, and paired t test or Wilcoxon test for within-group comparisons. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total knee arthroplasty
* Age ≥ 18 years
* ASA physical status classification I-III

Exclusion Criteria:

* Active infection
* Hematologic disease (e.g., leukemia, aplastic anemia)
* Autoimmune or chronic inflammatory disease
* Use of corticosteroids or immunosuppressive drugs
* Malignancy
* Acute trauma or sepsis
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective total knee arthroplasty at Elazig Fethi Sekin City Hospital, Department of Anesthesiology and Reanimation.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2025-09-22 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Change in Delta Neutrophil Index (DNI) | From baseline (preoperative) to 24 hours postoperative.
  Difference in DNI values measured preoperatively and postoperatively in patients undergoing total knee arthroplasty under spinal versus general anesthesia.

SECONDARY OUTCOMES:
Neutrophil Count | Preoperative to 24 hours postoperative.
  Absolute neutrophil count measured preoperatively and at 24 hours postoperatively.
Perioperative Complications | Intraoperative and during hospital stay (up to 7 days).
  Incidence of complications such as infection, bleeding, or cardiovascular events.
Operative Time | Intraoperative period.
  Duration of surgery recorded in minutes.
Lymphocyte Count | Preoperative to 24 hours postoperative.
  Absolute lymphocyte count measured preoperatively and at 24 hours postoperatively.
Neutrophil-to-Lymphocyte Ratio (NLR) | Preoperative to 24 hours postoperative.
  NLR calculated from complete blood count values preoperatively and at 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Şenol Karataş, Principal Investigator — Elazığ Fethi Sekin City Hospital, Department of Anesthesiology and Reanimation
Locations (1):
- University of Health Sciences, Elazığ Fethi Sekin City Hospital, Elâzığ, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is single-center, observational, and involves routine clinical laboratory results that are stored only in hospital records.

REFERENCES:
- [Background] Bozan MB, Yazar FM, Kale IT, Yuzbasioglu MF, Boran OF, Azak Bozan A. Delta Neutrophil Index and Neutrophil-to-Lymphocyte Ratio in the Differentiation of Thyroid Malignancy and Nodular Goiter. World J Surg. 2021 Feb;45(2):507-514. doi: 10.1007/s00268-020-05822-6. Epub 2020 Oct 16. PMID 33067685
- [Background] Nahm CH, Choi JW, Lee J. Delta neutrophil index in automated immature granulocyte counts for assessing disease severity of patients with sepsis. Ann Clin Lab Sci. 2008 Summer;38(3):241-6. PMID 18715852
- See also: Elazığ Fethi Sekin City Hospital, Department of Anesthesiology and Reanimation — https://elazigsehir.saglik.gov.tr/